CLINICAL TRIAL: NCT02592317
Title: Drug-drug Interaction Study to Evaluate the Effect of Multiple Doses of JNJ-56021927 on the Pharmacokinetics of Multiple Cytochrome P450 and Transporter Substrates in Subjects With Castration-Resistant Prostate Cancer
Brief Title: A Study to Evaluate the Effect of Multiple Doses of JNJ-56021927 on the Pharmacokinetics of Multiple Cytochrome P450 and Transporter Substrates in Participants With Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108072; 56021927PCR1020 (Other: Janssen Research & Development, LLC); 2015-003691-72 (EudraCT Number)
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: JNJ-56021927; Prostatic Neoplasms, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — Pioglitazone; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- JNJ 56021927 (Experimental): Participants will receive drug cocktail (comprising of midazolam [2 milligram {mg}], warfarin [10 mg], vitamin K (10 mg), omeprazole (40 mg), and fexofenadine [30 mg]) orally on Study Day 1 and 43 (Cycle 2 Day 1). On Study Day 8 and 50, pioglitazone 15 mg will be administered orally and on Study Day 9 and 51, rosuvastatin 10 mg will be administered orally. JNJ 56021927, 240 mg once daily will be administered on Study Day 15 up to disease progression, unacceptable toxicity, withdrawal of consent, lost to follow-up, the participant is no longer receiving clinical benefit in the opinion of the Investigator, the start of subsequent anticancer therapy, or the Sponsor ends the study.
  Interventions: Drug: JNJ 56021927; Drug: Drug Cocktail; Drug: Pioglitazone; Drug: Rosuvastatin

INTERVENTIONS:
Drug: JNJ 56021927 — JNJ 56021927 will be administered once daily orally in a dose of 240 mg from Study Day 15 up to disease progression, unacceptable toxicity, withdrawal of consent, lost to follow-up, the participant is no longer receiving clinical benefit in the opinion of the Investigator, the start of subsequent anticancer therapy, or the Sponsor ends the study.
Drug: Drug Cocktail — Drug cocktail comprise of midazolam (2 mg), warfarin (10 mg), vitamin K (10 mg), omeprazole (40 mg), and fexofenadine (30 mg) will be administered on Study Day 1 and 43.
Drug: Pioglitazone — Pioglitazone 15 mg will be administered orally on Study Day 8 and 50.
Drug: Rosuvastatin — Rosuvastatin 15 mg will be administered orally on Study Day 9 and 51.

SUMMARY:
The purpose of this study is to evaluate the effects of repeat dosing of JNJ-56021927 on the pharmacokinetics for single-dose multiple cytochrome P450 (CYP450) enzymes (CYP3A4, CYP2C9, CYP2C19, CYP2C8) and transporter (P-gp and BRCP) substrates in participants with castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label study in participants with CRPC. The study will consist of a Screening Phase to determine eligibility, a Pretreatment Phase, a Treatment Phase, and a Follow-up Phase. The study is designed to estimate the magnitude of the effects of JNJ-56021927 on the pharmacokinetics of probe substrates. In vitro studies have indicated that JNJ-56021927 and its active metabolite JNJ-56142060 (M3) have the potential to affect multiple cytochrome P450 (CYP) enzymes (CYP3A4, CYP2C9, CYP2C19, and CYP2C8) and drug transporters proteins (P-glycoprotein [P-gp] and breast cancer resistance protein [BRCP]) via inhibition or induction. In human hepatocytes, JNJ 56021927 and JNJ-56142060 (M3) were found to be inducers of CYP3A4. The induction of CYP3A4 suggests that JNJ-56021927 and M3 will induce other CYP isozymes and drug transporters (eg, CYP2C and P-gp via activation of pregnane X receptor). The study is designed to confirm the in vivo significance of these non-clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Adenocarcinoma of the prostate
* Participants with non-metastatic castration-resistant prostate cancer (NM-CRPC) or metastatic castration-resistant prostate cancer (mCRPC), who in the opinion of the investigator may benefit from treatment with JNJ-56021927
* Surgically or medically castrated, with testosterone levels of <50 nanogram per deciliter (ng/dL)
* If the participant is being treated with a gonadotropin-releasing hormone (GnRHa) (ie, participant who has not undergone bilateral orchiectomy), then this therapy must have been initiated at least 4 weeks prior to the Cycle 1 Day 1 visit and must be continued throughout the study
* Adequate bone marrow and organ function defined as: Hemoglobin (>=9.0 g/dL, independent of transfusion or growth factor support within the prior 7 days); Absolute neutrophil count (>=1000/mm^3 independent of growth factor support within the prior 7 days); Platelet count (>=75,000/mm^3 independent of transfusion or growth factor support within the prior 7 days); Serum albumin (>=3.0 g/dL); Serum creatinine (<=1.5*upper limit of normal (ULN) or calculated creatinine clearance >=50 mL/min/1.73m^2); Total bilirubin [<1.5*ULN (participants with Gilbert's Syndrome may be enrolled if the total bilirubin is <4 mg/dL with predominance of indirect bilirubin >=80% of total bilirubin]); Aspartate aminotransferase or alanine aminotransferase (<=3.0*ULN); Prothrombin time (PT) or partial thromboplastin time (PTT) or international normalized ratio (INR) (PT <=15 sec or INR <=1.2 PTT <=40 sec).

Exclusion Criteria:

* Known brain metastases
* Chemotherapy or immunotherapy for the treatment of prostate cancer within 4 weeks of the Study Day 15 (Cycle 1 Day 1) visit
* Prior treatment with enzalutamide within 8 weeks before first dose of drug probes
* Therapies that must be discontinued or substituted prior to study visit Day 1, or must be temporarily interrupted during the course of the study, include the following: a) Medications known to lower the seizure threshold within 4 weeks before Study Day 15 (Cycle 1 Day 1) and b) Medications known to induce or inhibit drug metabolizing enzymes (CYP3A4, CYP2C9, CYP2C19 and CYP2C8) or transporter proteins (P-gp, BRCP, OATP1B1, and OATPB3)
* Participant has known allergies, hypersensitivity, or intolerance to any of the study drugs/drug probes or excipients
* History of seizure or any condition that may predispose to seizure within 12 months prior to enrollment (Study Day 1); brain arteriovenous malformation; or intercranial masses such as schwannoma or meningioma that is causing edema or mass effect
* Participants with poor metabolizer genotype for CYP2C9 (*2, *3), or CYP2C19 (*2, *3, *4, *8)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1, 8, 9, 43, 50, and 51
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve. Cmax for Midazolam, S-warfarin, omeprazole, fexofenadine, pioglitazone, rosuvastatin will be assessed along with the metabolites of Midazolam, S-warfarin, omeprazole and pioglitazone.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Day 1, 8, 9, 43, 50, and 51
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time. AUC (0-last) for Midazolam, S-warfarin, omeprazole, fexofenadine, pioglitazone, rosuvastatin will be assessed along with the metabolites of Midazolam, S-warfarin, omeprazole and pioglitazone.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Day 1, 8, 9, 43, 50, and 51
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant. AUC[0-infinity]) for Midazolam, S-warfarin, omeprazole, fexofenadine, pioglitazone, rosuvastatin will be assessed along with the metabolites of Midazolam, S-warfarin, omeprazole and pioglitazone.

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Days 1, 8, 9, 43, 50, and 51
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration. Tmax for Midazolam, S-warfarin, omeprazole, fexofenadine, pioglitazone, rosuvastatin will be assessed along with the metabolites of Midazolam, S-warfarin, omeprazole and pioglitazone.
Elimination Rate Constant (Lambda[z]) | Day 1, 8, 9, 43, 50, and 51
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve. Lambda[z]) for midazolam, S-warfarin, omeprazole, fexofenadine, pioglitazone, rosuvastatin will be assessed along with the metabolites of Midazolam, S-warfarin, omeprazole and pioglitazone.
Elimination Half-Life (t1/2) | Days 1, 8, 9, 43, 50, and 51
  The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z). t1/2 for Midazolam, S-warfarin, omeprazole, fexofenadine, pioglitazone, rosuvastatin will be assessed along with the metabolites of Midazolam, S-warfarin, omeprazole and pioglitazone.
Apparent Clearance (CL/F) | Days 1, 8, 9, 43, 50, and 51
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F for Midazolam, S-warfarin, omeprazole, fexofenadine, pioglitazone, rosuvastatin will be assessed along with the metabolites of Midazolam, S-warfarin, omeprazole and pioglitazone.
Maximum Observed Plasma Concentration (Cmax) for JNJ-56021927 | Day 43
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) for JNJ-56021927 | Day 43
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24]) | Day 43
  The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours.
Trough Plasma Concentration (Ctrough) | Day 43, 50 and 51
  The (Ctrough) is the plasma concentration before dosing or at the end of the dosing interval of any dose other than the first dose in a multiple dosing regimen.
Number of Participants with Adverse Events | Up to 6 years 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (3):
- Chisinau, Moldova
- Spain (2):
  - Barcelona
  - Seville